CLINICAL TRIAL: NCT06514300
Title: MYO-SLD : a Prospective Study to Determine the Phenotype of Muscle Fat Accumulation in a Cohort of Patients With SLD as to Confirm the Association Between Muscle Composition and Texture and the Phenotype of Liver Disease
Brief Title: Investigating Myosteatosis in Steatotic Liver Diseases
Acronym: MYO-SLD
Status: Enrolling by invitation | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other); Concerted Research Action (Unknown)
Responsible Party: Sponsor
Other Study IDs: ST-IR-01 - MYO-SLD
Record Dates: First submitted 2024-06-27; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Alcohol-related Liver Disease; Metabolic Dysfunction Associated Steatotic Liver Disease; Steatotic Liver Disease of Mixed Origin (MetALD); Steatotic Liver Diseases; Myosteatosis; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Liver Histology
Keywords: myosteatosis; steatotic liver disease; metabolic dysfunction-associated steatotic liver disease; alcohol-related liver disease; MetALD; magnetic resonance imaging; magnetic resonance spectroscopy; liver biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * liver biopsy
  * serum/plasma samples
  * urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MASLD patients: patients presenting with liver steatosis and at least one cardiometabolic criteria.
- ALD patients: patients presenting with liver steatosis secondary to an excessive consumption of alcoholic beverages and with no cardiometabolic criteria.
- MetALD patients: patients presenting with liver steatosis, at least one cardiometabolic criteria and an excessive consumption of alcohol beverages.

SUMMARY:
Steatotic liver diseases (SLD) are the most common chronic liver diseases worldwide. SLD are defined by an excessive liver lipid content (steatosis) of more than 5% of the total liver weight and includes 3 clinical entities : metabolic dysfunction-associated steatotic liver disease (MASLD), alcohol-related liver disease (ALD) and a mixed entity combining the two settings referred as MetALD. SLD are associated to extra-hepatic complications such as cardiovascular diseases, insulin resistance or muscle changes. Among the latter, myosteatosis, defined by an excessive muscle fat content, has been reported as a muscle change in MASLD occuring even in non-cirrhotic stages. Investigators will explore these muscle changes in SLD patients according to the severity of the underneath liver disease.

DETAILED DESCRIPTION:
This project investigates the correlation between liver and muscle phenotypes assessed in a cohort of all 3 SLD subgroups (MASLD, ALD and MetALD). If a severe form of SLD is suspected based on a severely increased liver elasticity, assessed by transient elastography, participants undergo a liver biopsy, liver and muscle magnetic resonance imaging. Eating habits and physical activity level are recorded using the 24 hour-recall and international physical activity questionnaire. Psychological disorders are also screened using dedicated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age between18 to 75 years
* Presence of hepatic steatosis, suggested by a controlled attenuation parameter (CAP) ≥ 252 dB/m on elastometry and elevated transaminases (ALT ≥ 25 or 33 IU/L in women or men respectively)
* Presence of overweight (BMI > 25 kg/m²), obesity (BMI > 30 kg/m²), metabolic syndrome, prediabetes or type 2 diabetes. Metabolic syndrome is defined by int ernational Diabetes Federation as follows : waist circumference ≥ 94/80cm for men/women with ≥ 2 other criteria: arterial pressure ≥ 130/85 mmHg or treatment for hypertension, fasting glucose ≥ 130/85 mmHg or treatment for hypertension, serum triglycerides > 150 mg/dl or treatment for dyslipidemia, HDL cholesterol < 40/50 mg/dl for men/women or treatment for dyslipidemia.

Exclusion Criteria:

* Liver disease from other causes (alcohol, active viral chronic hepatitis B or C, Wilson's disease, autoimmune hepatitis, alpha1-anti-trypsin deficiency,...)
* Heavy consumption of alcoholic beverages, i.e. > 140 g or 210 g of ethanol in women or men respectively).
* Intravenous drug use
* HbA1C > 10%
* Decompensated cirrhosis (presence of ascites, bilirubin level > 1.2 mg/dL in a patient without Gilbert's syndrome, albumin level < 35 g/L)
* Pregnancy
* Use of drugs that may cause steatosis (methotrexate, amiodarone, tamoxifen, oral corticosteroids) currently or in the last 3 months
* Change in treatment of hyperglycaemia (dose or medication) in the last 3 months
* Change in body weight >5% in the last 3 months
* Active cancer
* End stage renal disease or dialysis
* Type 1 diabetes or secondary diabetes
* Digestive malabsorption
* Untreated thyroid disease
* Taking a treatment under study or approved for NASH (semaglutide, lanifibranor, obeticholic acid).
* Musculoskeletal disorders, neuromuscular or inflammatory diseases such as connective tissue diseases, myositis and vasculitis that have musculoskeletal manifestations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is intended for patients with steatotic liver diseases SLD) characterized by an excessive liver lipid content higher than 5% (steatosis). SLD include 3 clinical entities with specific diagnostic criteria previously defined (Rinella MC, et al. J Hepatol. 2023) : metabolic dysfunction-associated steatotic liver disease, highly related to overweight, obesity and type 2 diabetes; alcohol-related liver disease, secondary to an excessive alcohol beverages consumption; and a third mixed entity combining both conditions called MetALD. All SLD patients will be recruited in this project to investigate if muscle phenotype is specifically related to one type of SLD.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
correlation between muscle mass and fat content and liver histological features of SLD | MRI and liver biopsy are performed at Day 1
  muscle mass and fat content will be assessed by magnetic resonance imaging and spectroscopy. Liver phenotype will be histologically assessed by 3 blinded pathologists and computer-assisted morphometry.

SECONDARY OUTCOMES:
liver molecular mechanisms involved in myosteatosis pathogenesis | liver samples are collected during the biopsy
  mRNA extraction and sequencing from liver tissue samples collected during liver biopsy to assess the transcriptomic pattern correlating with muscle fat assessed by MRI.
impact of muscle fat content on muscle function | muscle function tests are performed 1-week after the biopsy/MRI (Day 7)
  investigators assess the correlation between muscle fat assessed by MRI and muscle function assessed by several tests.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Lanthier, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linge J, Nasr P, Sanyal AJ, Dahlqvist Leinhard O, Ekstedt M. Adverse muscle composition is a significant risk factor for all-cause mortality in NAFLD. JHEP Rep. 2022 Dec 24;5(3):100663. doi: 10.1016/j.jhepr.2022.100663. eCollection 2023 Mar. PMID 36818816
- [Background] Ong JP, Pitts A, Younossi ZM. Increased overall mortality and liver-related mortality in non-alcoholic fatty liver disease. J Hepatol. 2008 Oct;49(4):608-12. doi: 10.1016/j.jhep.2008.06.018. Epub 2008 Jul 9. PMID 18682312
- [Background] Singal AK, Mathurin P. Diagnosis and Treatment of Alcohol-Associated Liver Disease: A Review. JAMA. 2021 Jul 13;326(2):165-176. doi: 10.1001/jama.2021.7683. PMID 34255003
- [Background] Rinella ME, Lazarus JV, Ratziu V, Francque SM, Sanyal AJ, Kanwal F, Romero D, Abdelmalek MF, Anstee QM, Arab JP, Arrese M, Bataller R, Beuers U, Boursier J, Bugianesi E, Byrne CD, Castro Narro GE, Chowdhury A, Cortez-Pinto H, Cryer DR, Cusi K, El-Kassas M, Klein S, Eskridge W, Fan J, Gawrieh S, Guy CD, Harrison SA, Kim SU, Koot BG, Korenjak M, Kowdley KV, Lacaille F, Loomba R, Mitchell-Thain R, Morgan TR, Powell EE, Roden M, Romero-Gomez M, Silva M, Singh SP, Sookoian SC, Spearman CW, Tiniakos D, Valenti L, Vos MB, Wong VW, Xanthakos S, Yilmaz Y, Younossi Z, Hobbs A, Villota-Rivas M, Newsome PN; NAFLD Nomenclature consensus group. A multisociety Delphi consensus statement on new fatty liver disease nomenclature. J Hepatol. 2023 Dec;79(6):1542-1556. doi: 10.1016/j.jhep.2023.06.003. Epub 2023 Jun 24. PMID 37364790
- [Background] Nachit M, Lanthier N, Rodriguez J, Neyrinck AM, Cani PD, Bindels LB, Hiel S, Pachikian BD, Trefois P, Thissen JP, Delzenne NM. A dynamic association between myosteatosis and liver stiffness: Results from a prospective interventional study in obese patients. JHEP Rep. 2021 Jun 15;3(4):100323. doi: 10.1016/j.jhepr.2021.100323. eCollection 2021 Aug. PMID 34355155
- [Background] Nachit M, Kwanten WJ, Thissen JP, Op De Beeck B, Van Gaal L, Vonghia L, Verrijken A, Driessen A, Horsmans Y, Francque S, Leclercq IA. Muscle fat content is strongly associated with NASH: A longitudinal study in patients with morbid obesity. J Hepatol. 2021 Aug;75(2):292-301. doi: 10.1016/j.jhep.2021.02.037. Epub 2021 Apr 15. PMID 33865909
- [Background] Henin G, Loumaye A, Leclercq IA, Lanthier N. Myosteatosis: Diagnosis, pathophysiology and consequences in metabolic dysfunction-associated steatotic liver disease. JHEP Rep. 2023 Nov 14;6(2):100963. doi: 10.1016/j.jhepr.2023.100963. eCollection 2024 Feb. PMID 38322420
- [Derived] Henin G, Goffaux A, Declerck S, Andre-Dumont S, Pendeville E, Valet M, Lejeune T, Dahlqvist G, Loumaye A, Schnabl B, Starkel P, Lanthier N. Non-Cirrhotic Steatotic Liver Disease is Associated With Impaired Muscle Function: A Cross-Sectional Study. JCSM Commun. 2025 Jul-Dec;8(2):e70012. doi: 10.1002/rco2.70012. Epub 2025 Oct 7. PMID 41127673